CLINICAL TRIAL: NCT07090239
Title: French Translation of the Self-administered Questionnaire The Female Sexual Distress Scale-Revised
Brief Title: French Translation of The Female Sexual Distress Scale-Revised
Acronym: f-FSDS-R
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0396 - f-FSDS-R
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-03

CONDITIONS: The Translation of a Screening Tool

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Two independent teams (Brest and Nice) each produce a forward translation from English to French. The translations are compared, and discrepancies are discussed with the translation coordinator, the second translator, and the scientific lead to produce a unified preliminary French version (Version 1), including the response options.

Version 1 is then back-translated into English by an English-speaking linguist and a French physician whose native language is English, without access to the original questionnaire, in order to detect potential translation issues. The team then holds a discussion to compare the original English version, the French Version 1, and the back-translations, resulting in the development of Version 2.

Version 2 is tested with a representative sample of patients using a paper questionnaire, which includes two follow-up questions after each item to assess comprehension and identify potential difficulties. The team analyzes the responses, and if comprehension issues are identified, they organize further discussions with the translators and back-translators to revise the items concerned. The revised items are then re-tested with patients, including those who have and have not reported difficulties, to ensure that the final version is clear and understandable for all.

the investigators conduct prospective recruitment after verifying the inclusion and exclusion criteria.

Inclusion criteria:

Adult patient Affiliation with a social security scheme

Exclusion criteria:

Patients under legal protection (guardianship, curatorship, etc.) Refusal to participate Patients with difficulties understanding the French language Patients consulting in the adult or gynecological emergency department, or accompanying another person, are informed about the possibility of completing a questionnaire.

The participants informed that their data will be recorded for the purpose of practice evaluation and results analysis in an anonymous and confidential manner, using the information sheet provided for the study. The participants free to refuse participation without any impact on their care.

Patients receive complete and clear information regarding the objectives of the study, their right to refuse participation, and their right to withdraw at any time. All this information appears on the information and non-opposition form provided to each patient. Participation is noted in the patient's medical record.

Administration procedures:

The questionnaire is distributed in the waiting area and is self-administered by the patient. Once consent is given, the patient completes the questionnaire independently.

Follow-up:

The estimated participation time is approximately 10 minutes, corresponding to the time required to complete the questionnaire. Patients may be contacted again if necessary to re-test reformulated items, including those who reported comprehension difficulties and others who did not.

The inclusion period lasts 6 months. The individual participation time is 10 minutes. The total duration of the prospective study (inclusion + follow-up) is 8 months.

The overall study timeline (including data entry and management of non-opposition forms) is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* affiliated to a social security scheme

Exclusion Criteria:

* Patients under judicial protection (guardianship, curatorship, ...)
* Refusal to participate
* Patient having difficulties understanding the French language.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients consulting in gynecology, obstetrics and adult emergencies, as well as those accompanying a third party.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the item-by-item response rate to the paper-based questionnaire, assessing the acceptability and feasibility of the French version of the FSDS-R in the target population. | from March to September 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement